CLINICAL TRIAL: NCT02374125
Title: Effectiveness of Teres Major Muscle Specific Treatment in Patients Diagnosed With Subacromial Impingement Syndrome
Brief Title: Teres Major Muscle and Subacromial Impingement Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P14/033
Record Dates: First submitted 2015-02-10; First posted 2015-02-27 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Trigger Points in Teres Major Muscle; Subacromial Impingement Syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fibrolysis Group (Experimental): Actual Diacutaneous Fibrolysis and protocolized physiotherapy
  Interventions: Device: Diacutaneous Fibrolysis; Other: Protocolized physiotherapy
- Pressure Group (Experimental): Trigger Point Pressure Release and protocolized physiotherapy
  Interventions: Other: Trigger Point Pressure Release; Other: Protocolized physiotherapy
- Control Group (Active Comparator): Protocolized physiotherapy
  Interventions: Other: Protocolized physiotherapy

INTERVENTIONS:
Device: Diacutaneous Fibrolysis — Applied only around teres major muscle.
  Arms: Fibrolysis Group
Other: Trigger Point Pressure Release — Applied only in teres major muscle trigger points.
  Arms: Pressure Group
Other: Protocolized physiotherapy — Exercises, TENS and cryotherapy

SUMMARY:
There is not a clear understanding of the origin of symptoms perceived by patients with impingement of the soft tissue structures of the subacromial space. Tendinopathy, tendon rupture or other pathologies, are present in asymptomatic subjects and subjects with symptoms and structural integrity can also be found.

Patients diagnosed with subacromial impingement syndrome frequently have myofascial trigger points in the teres major muscle. Travell and Simons reported that the symptoms caused by trigger points in this muscle are similar to those experienced by patients diagnosed with impingement syndrome, but a literature search provides few results regarding relationship between subacromial impingement syndrome and presence of myofascial trigger points in the teres major muscle.

This study aims to provide evidence of the results that can be obtained with a specific approach of teres mayor muscle by two manual techniques, Trigger Point Pressure Release and Diacutaneous Fibrolysis, in subjects with subacromial impingement syndrome, a condition that still representing both a diagnostic and therapeutic challenge. Secondary objective is to compare the outcomes between both techniques to select for each patient the most appropriate to their needs and characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and over
* Clinical diagnosis of Subacromial Impingement Syndrome.
* Detectable trigger points in teres major muscle.
* Sign informed consent form.

Exclusion Criteria:

* Diacutaneous Fibrolysis contraindications
* Previous shoulder surgery (<1year)
* Language barriers or cognitive issues that limit their ability to provide informed consent and participate in research.
* Patients with a pending litigation or court claim.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change in Pain intensity (Using a VAS) | Change from baseline to 3 weeks.
  Using a VAS
Change in Functional capacity (Abbreviated Constant-Murley score) | Change from baseline to 3 weeks.
  Abbreviated Constant-Murley score

SECONDARY OUTCOMES:
Change in Active Range of Motion | Change from baseline to 3 weeks.
  Flexion, extension, abduction, external rotation and internal rotation
Patient perception of change (Global Rating of Change scale) | 3 weeks after recruitment
  Global Rating of Change scale

CONTACTS AND LOCATIONS:
Overall Officials: Martín Barra, Principal Investigator — Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Locations (1):
- Catalan Health Institut. Sant Ildefons Rehabilitation Service, Cornellà de Llobregat, Barcelona, Spain